CLINICAL TRIAL: NCT04242810
Title: Effects of rTMS on Human Brain Activity Measured With fMRI
Brief Title: Effects of rTMS on Human Brain Activity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started enrollment due to COVID-19 closures
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00102980
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Repetitive Transcranial Magnetic Stimulation (rTMS)
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): rTMS applied over memory task-based brain target
  Interventions: Device: rTMS; Procedure: MRI scan
- Sham rTMS (Placebo Comparator): Sham rTMS applied over memory task-based brain target
  Interventions: Device: Sham rTMS; Procedure: MRI scan

INTERVENTIONS:
Device: rTMS — TMS will be applied over task-based target at an intensity up of 130% rMT. The optimal coil placement during stimulation will be guided using the BrainSight neuronavigation system.
  Arms: Active rTMS
Device: Sham rTMS — An electrical sham coil that produces the same auditory and somatosensory stimulations, without a significant magnetic field, will be used as an active control.
  Arms: Sham rTMS
Procedure: MRI scan — Participants will undergo an MRI scan directly after rTMS stimulation that will last less than 120 minutes. During the scan, subjects will encode and retrieve object pictures.

SUMMARY:
The purpose of this study is to investigate how repetitive transcranial magnetic stimulation (rTMS) affects brain networks measured by functional magnetic resonance imaging (fMRI).

Participants will undergo a screening that includes a psychiatric and medical history screening, TMS and MRI safety screening, and urine screening. If participants pass the screening procedure, they will be introduced to transcranial magnetic stimulation (TMS), magnetic resonance imaging (MRI), and a task that involves viewing words, sentences, or pictures. There will be up to seven visits and each visit will take less than 3 hours.

MRI can be dangerous for people that have medical devices, metal objects, or metal debris in their bodies. TMS procedures are associated with a very low risk of seizures, "muscle-tension" type headache, ear damage, numbness of the face, fainting, dizziness, memory impairment, trouble concentrating, and acute mood changes. This study will use only levels of TMS that are within safety guidelines. There is also a risk of potential loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Age restrictions: between 18-35 years old
* Use of effective method of birth control for women of childbearing capacity.
* Willing to provide informed consent.

Exclusion Criteria:

* Current or recent (within the past 6 months) substance abuse or dependence, excluding nicotine and caffeine (urine test)
* Current serious medical illness (self-report)
* History of seizure except those therapeutically induced by ECT (childhood febrile seizures are acceptable and these subjects may be included in the study), history of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion, devices that may be affected by rTMS or MRI (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Subjects are unable or unwilling to give informed consent
* Diagnosed any Axis I DSM-IV disorder (MINI, DSM-IV)

Subjects with a clinically defined neurological disorder including, but not limited to:

* Any condition likely to be associated with increased intracranial pressure
* Space occupying brain lesion.
* History of stroke.
* Transient ischemic attack within two years.
* Cerebral aneurysm.
* Dementia.
* Parkinson's disease.
* Huntington's disease.
* Multiple sclerosis.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold
* Subjects with cochlear implants
* Subjects not willing to tolerate the confinement associated with being in the MRI scanner
* Women who are pregnant or breast-feeding (urine test)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of a rTMS session on the performance for a memory task, as measured by accuracy (in percentage of correct responses) | up to 1 month
An effect of a rTMS session on the performance for a memory task, as measured by reaction time (in ms) | Time frame: up to 1 month
An effect of a rTMS session on fMRI brain representation for a memory task, as measured by BOLD signal | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cabeza, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No